CLINICAL TRIAL: NCT03137095
Title: Longitudinal Pilot Mechanistic Study of the Effects of Chemotherapy on Cognitive Function in Breast Cancer Patients and Non-Cancer Control Participants - Optional Sub-Study: Research Brain MRI
Brief Title: Effects of Chemotherapy on Cognitive Function in Breast Cancer Patients & Non-Cancer Control Subjects With Optional Sub-Study Research Brain MRI
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michelle Janelsins, PhD, MPH, Assistant Professor, University of Rochester
Other Study IDs: 54027
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cancer Related Cognitive Difficulties; Breast Cancer Female
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Patient Participants: Female breast cancer patients receiving chemotherapy
  Interventions: Other: Cognitive testing; Other: Research Brain MRI
- Healthy, age-matched, female participants: Healthy, female, age-matched participants
  Interventions: Other: Cognitive testing; Other: Research Brain MRI

INTERVENTIONS:
Other: Cognitive testing — computerized and paper-based cognitive tests that assess memory, executive function, processing speed and concentration performed at Assessments 1, 3, 4.5 & 5.
Other: Research Brain MRI — Optional sub-study participation includes undergoing research brain MRI to obtain structural and functional brain images at Assessment 4.5 and 6.

SUMMARY:
Study is enrolling newly diagnosed breast cancer patients about to start chemotherapy and age-matched control participants. The investigator is trying to better understand the prevalence of cognitive difficulties in cancer patients receiving chemotherapy compared to the general population as well as what biological mechanisms may play a role in the development of these difficulties. Patients will be asked to complete six assessments over the course of approximately 5 months. Assessments 1,3, 4.5 and 5 include computerized and paper and pencil cognitive testing as well as blood draws. Assessments 2 and 4 only involve the collection of a blood sample. An optional sub study is offered after Assessment 1. It involves a research brain MRI at Assessment 4.5 and cognitive testing and another research brain MRI at Assessment 6.

ELIGIBILITY:
Inclusion Criteria, Breast Cancer Patient Participants:

* Females with a diagnosis of invasive non-metastatic breast cancer (stage I-IIIC)
* Scheduled to begin a course of chemotherapy with Adriamycin and Cytoxan
* Chemotherapy naïve
* Able to speak and read English
* 21 years or older
* Give written informed consent

Exclusion Criteria, Breast Cancer Patient Participants:

* Must not be currently hospitalized or have been hospitalized within the last year for a psychiatric illness
* Must not be diagnosed with a neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease)
* Must not have any Central Nervous System disease (e.g., movement disorder, multiple sclerosis)
* Subjects could have had a TIA (transient ischemic attack) or stroke in the past if the TIA or stroke was greater than 1 year ago and the subject does not have any remaining symptoms
* Must not be scheduled to receive concurrent radiation treatment while receiving chemotherapy.
* Must not be colorblind

Inclusion Criteria, Control Participants:

* Must be female and within 5 years of the age of the subject receiving chemotherapy
* Able to speak and read English
* Give written informed consent
* 21 years or older

Exclusion Criteria, Control Participants:

* Must not be currently hospitalized or have been hospitalized within the last year for a psychiatric illness
* Must not be diagnosed with a neurodegenerative disease (e.g. Alzheimer's disease, Parkinson's disease)
* Must not have Central Nervous System disease (e.g., movement disorder, multiple sclerosis)
* Subjects could have had a TIA (transient ischemic attack) or stroke in the past if the TIA or stroke was greater than 1 year ago and the subject does not have any remaining symptoms
* Must not have been diagnosed with cancer or previously have received chemotherapy
* Must not be colorblind

For optional sub-study: MR safety assessed via Rochester Center for Brain Imaging Magnetic Resonance (MR) Safety Screening Form to confirm eligibility to participate

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female breast cancer patients with a diagnosis of invasive non-metastatic breast cancer (stage I -IIIC) and age-matched, health female participants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function (memory, concentration, attentiveness) will be assessed by computerized cognitive assessments and associated with inflammation and neurotoxicity markers | During chemotherapy and 1 month post-chemotherapy; Approximately 3 - 5 months
  Change scores from baseline will be computed for each cognitive measure as well as each mechanistic marker

OTHER OUTCOMES:
Research Brain MRI | After 4 cycles Adriamycin/Cytoxan (each cycle of AC is 14 days) and within 1 month post additional chemotherapy treatment
  MRI brain imaging to obtain structural and connectivity data via fMRI (brain function), T1MRI (brain structure) and DTI (white matter related microstructure in brain) to determine if there are changes within the brain related to cognitive performance, symptoms, immune and other biologic factors

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C. Janelsins, Ph.D.,M.P.H., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States